CLINICAL TRIAL: NCT03678597
Title: Latrunculin B Supplementation to ICSI Handling Medium
Brief Title: Supplementing Intracytoplasmic Sperm Injection Handling Medium With Latrunculin B ( ICSI-LB)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibn Sina Hospital (Other Government)
Responsible Party: Principal Investigator, Muhammad Fawzy, IVF Lab Director, Ibn Sina Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IbnSinaIVF-ICSI-LB
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — latrunculin B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Handling Medium Supplemented with Latrunculin B (Experimental)
  Interventions: Other: Medium Supplemented with Latrunculin B
- handling Medium as it is. (No Intervention)

INTERVENTIONS:
Other: Medium Supplemented with Latrunculin B — A medium with in-house supplementation of Latrunculin B to decrease oocyte degeneration after ICSI and improve the survival rate
  Arms: Handling Medium Supplemented with Latrunculin B

SUMMARY:
Vienna Consensus has identified 10% damage rate after ICSI as a competency value. Despite the highest quality embryologists doing ICSI, degeneration sometimes occurs due to oocyte factors such as the fragile membrane, etc. Latrunculin B serves to facilitate spindle or pronuclear transfer procedures helping to reduce the damage rate with no harm reported. Using Latrunculin B during ICSI could serve to rescue some oocytes from the degeneration allowing for more chances of viable zygotes,

ELIGIBILITY:
Inclusion Criteria:

* All ICSI cycles

Exclusion Criteria:

-

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
oocyte survival rate after ICSI | 6 days of culture

SECONDARY OUTCOMES:
Fertilisation rate | 6 days of culture
Rates of blastocyst formation and quality | 6 days of culture
  Number of formed and high-quality blastocysts per fertilized oocytes
Clinical pregnancy rate | three months
Implantation rate | 7 weeks
Ongoing pregnancy rate | 12 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- Egypt (3):
  - Qena Fertility Center, Qina, Qena Governorate
  - Banon Assiut, Asyut
  - IbnSina IVF Center, IbnSina Hospital, Sohag